CLINICAL TRIAL: NCT00596375
Title: Lidocaine Lubricant Use as an Anesthetic Agent in Emergency Room Urethral Catheterization
Brief Title: Lidocaine Lubricant in Pediatric Urethral Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Emory University (Other)
Responsible Party: Michael Greenwald, MD, Children's Healthcare of Atlanta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 06693
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-12

CONDITIONS: Fevers; Pain
Keywords: Lidocaine; Infant; Urinary Catheterization; Emergency Medicine; Analgesia
MeSH Terms: conditions — Fever; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Routine Care Group (No Intervention): The routine care group will help us to quantify the routine amount of distress associated with catheterization.
- Lidocaine Group (Experimental): A experimental group will include patients who will have 2% Lidocaine instilled into the urethra prior to catheterization. This group of subjects receiving routine care plus Lidocaine, will be evaluated during each of the four phases of the intervention.
  Interventions: Drug: Lidocaine Lubricant
- Instillation (Experimental): This group will undergo catheterization utilizing routine care plus lubricant jelly instilled into the urethra. This placebo group will aid in discerning the effects of instillation into the urethra on pain and associated distress.
  Interventions: Procedure: Lubricant Instillation

INTERVENTIONS:
Procedure: Lubricant Instillation — Lubricant jelly instilled in urethra prior to catheterization
  Arms: Instillation
Drug: Lidocaine Lubricant — 2% Lidocaine lubricant instillation prior to urethral catheterization
  Arms: Lidocaine Group

SUMMARY:
In Emergency Departments (ED) across the nation there is renewed interest in finding ways to alleviate the pain and discomfort associated with many of the procedures that children must undergo. In a policy by the American Academy of Pediatrics, a nationally recognized advocate for children, physicians are urged to advocate for child-specific research in pain management and the effective use of pain medication to ensure compassionate and competent management of pain. (AAP Statement, 2001) Pediatric urethral catheterizations are one such procedure in which children experience significant pain.(11) In present care, children over 2 months of age do not routinely receive intervention for urethral catheterization related anxiety and pain, and, anecdotal reports suggest that most require physical restraint to complete the procedure. Lidocaine is an anesthetic agent that provides relief from pain during many commonly performed ED procedures. Intraurethral Lidocaine has been shown to decrease pain associated with urethral catheter placement in cystograms, however, Lidocaine is not routinely used for urethral catheterizations in the CHOA ED.

This study aims to investigate the potential use of Lidocaine as an anesthetic agent during urethral catheterization of children. Recently, two specific studies were performed investigating the use of Lidocaine to decrease discomfort associated with urethral catheterization. Using the strengths of both previously published studies, our study will use Lidocaine both topically and instilled into the urethra. Investigators plan to perform a prospective three-arm double-blinded randomized clinical trial investigating the effectiveness of Lidocaine jelly as a analgesic when used as a lubricant for urinary catheterization. Investigators aim to demonstrate that Lidocaine used as a lubricant anesthetic for urethral catheterization will provide a safe, time-efficient, and relatively easy way to decrease pediatric pain in the emergency department setting.

DETAILED DESCRIPTION:
In Emergency Departments (ED) across the nation there is renewed interest in finding ways to alleviate the pain and discomfort associated with many of the procedures that children must undergo. Children's memory and reaction to negative experiences in the care of medical professionals has led to many changes in procedural pain management (4). One noxious procedure that continues to be performed in the ED without the use of anesthetic agents is urethral catheterization (11). In a policy by the American Academy of Pediatrics, a nationally recognized advocate for children, physicians are urged to advocate for child-specific research in pain management and the effective use of pain medication to ensure compassionate and competent management of pain. (AAP Statement, 2001)

Pediatric urethral catheterizations are one such procedure in which children experience significant pain. (11) The Children's Healthcare of Atlanta (CHOA) ED at Egleston performs an average of greater than 150 pediatric urethral catheterizations per month. This procedure is performed in most cases where children under 6 months of age present with unexplained fever. Also, divisional guidelines call for urethral catheterization for urinanalysis and urine culture on all uncircumcised boys under the age of 1 and all girls under the age of 2 who present with unexplained temperature above 39.5 degrees. In a previous Friends funded clinical trial, ED investigators studied sucrose use in children under 2 months of age which was shown to decrease urethral catheterization discomfort. As such, this has become routine care in the ED. (REF; for a review of sucrose for pediatric pain, see 6) In present care, children over 2 months of age do not routinely receive intervention for urethral catheterization related anxiety and pain, and, anecdotal reports suggest that most require physical restraint to complete the procedure.

Lidocaine is an anesthetic agent that provides relief from pain during many commonly performed ED procedures. Examples of present Lidocaine use in the ED are laceration repair, abscess drainage, and lumbar puncture. Given the anxiety, discomfort, and pain associated with urethral catheterizations (1, 2, 3, 4), Lidocaine has begun to be used clinically in this arena. Intraurethral Lidocaine has been shown to decrease pain associated with urethral catheter placement in cystograms, however, Lidocaine is not routinely used for catheter placement to obtain urine in the CHOA ED.

Recently, two specific studies were performed investigating the use of Lidocaine to decrease discomfort associated with urethral catheterization. The first published study supports the use of intraurethral Lidocaine for catheterization.(5) In this investigation, Lidocaine was repeatedly instilled into the urethra of ten 4- to 11-year-old patients for approximately 10 minutes prior to a scheduled cystogram. Patients in this study indicated significantly less pain with Lidocaine as a lubricant when compared to those who received sterile lubricant jelly. However, the placement of a catheter for cystogram requires the catheter to be in place for the duration of the procedure (10 to 15 minutes); whereas catheterization in the ED for urinalysis and urine culture requires catheter placement for a much shorter period of time. The second study, which compared Lidocaine to lubricant jelly used as a topical anesthetic prior to catheterization, found that preverbal patients experienced the same discomfort with or without Lidocaine when evaluated using Face-Legs-Activity-Cry-Consolability (FLACC) scoring.(11) Authors attempted to investigate Lidocaine topically placed at the urethral meatus to provide relief. Although the investigators did not achieve their goal of pain reduction using Lidocaine topically, they did find that the incidence of positive urine culture was similar in both the Lidocaine and placebo groups. Using the strengths of both previously published studies, our study will use Lidocaine both topically and instilled into the urethra.

Medical care professionals are increasing their attention to pain and comfort measures for children undergoing painful procedures in the ED. Pediatric urethral catheterization is one such area that remains unaddressed. The use of Lidocaine as an anesthetic in common ED procedures is well known. Investigation of Lidocaine use as an anesthetic lubricant has been reported twice previously in pediatric literature with contradicting results. After critical appraisal of these studies, our investigators conclude that additional investigation is warranted with the following characteristics: Lidocaine should be placed both topically and instilled into the urethra; Lidocaine should be compared to both routine care and placebo; methodology should include blinded observations; methodology should evaluate pain response utilizing numerous validated tools; and urine should be monitored to evaluate the biological effects of Lidocaine on urine culture results. Investigators aim to demonstrate that Lidocaine used as a lubricant anesthetic for urethral catheterization will provide a safe, time-efficient, and relatively easy way to decrease pediatric pain in the emergency department setting.

Specific Aims & Hypotheses

SA1: To study the potential use of Lidocaine as an anesthetic agent during urethral catheterization of children presenting to Pediatric Emergency Department.

H1: The use of Lidocaine jelly as a lubricant in urethral catheterizations in pediatric ED patients significantly decreases distress associated with this procedure.

SA2: To determine the average Lidocaine concentration present in urine obtained with Lidocaine jelly used as lubricant during urinary catheterization.

H2: Urine Lidocaine concentrations associated with routine urethral catheterization utilizing intraurethral Lidocaine installation will not approach known bacterial growth-limiting levels.

ELIGIBILITY:
Inclusion Criteria:

* Febrile patients aged 2 months to 2 years receiving urethral catheterization to obtain sterile urine for microbiologic and chemistry testing will be eligible to participate. Our study will be limited to children presenting with fever secondary to an unknown source, as ED triage protocol requires the administration of non-steroidal analgesic to treat fever.

Exclusion Criteria:

* The physician determines the patient is in need of immediate treatment or catheterization
* Patients have a history of genitourinary abnormalities
* Patients have had a previous catheterization
* Primary caregiver has limited English proficiency
* Patients with a history of genitourinary abnormalities
* Patients with history of prior catheterization are excluded from enrollment

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2006-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Modified Behavior Pain Scale | Procedure (approx. 6 minutes)

SECONDARY OUTCOMES:
Lidocaine Concentration | Procedure (approx. 6 minutes)
Visual Analog Scale | Procedure (approx. 6 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Greenwald, MD, Principal Investigator — Children's Healthcare of Atlanta; Patrick P Mularoni, MD, Study Director — Johns Hopkins All Children's Hospital
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States